CLINICAL TRIAL: NCT01774175
Title: A Randomised Controlled Trial of a 2 Litre Polyethylene Glycol Solution + Ascorbic Acid Versus Sodium Picosulphate + Magnesium Citrate Solution for Bowel Cleansing Prior to Colonoscopy
Brief Title: Comparison Between Coolprep and Picolyte for Bowel Cleansing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Chung Jun Won, Professor, Gachon University Gil Medical Center
Other Study IDs: COOLPREPICOLYTE
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Stasis; Colon
Keywords: Bowel preparation; PEG with ascorbic acid; Picosulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Coolprep: A total of 2L A : NaCl 5.382g KCl 2.03g Sodium sulfate 15g Polyethylene glycol 3350 200.0g B : Ascorbic acid 9.4g Sodium ascorbate 11.8g
- Picolyte: Sodium picosulfate 30.0mg Magnesium citrate 10.5g + 36.0g

SUMMARY:
The investigators will compare with PEG+ascorbic acid and picosulfate+magnesium citrate about bowel preparation, patient's satisfaction, side effects to identify effectiveness of new bowel preparation drug.

DETAILED DESCRIPTION:
The investigators can find easily colon cancer and poly by colonoscopy, but bowel preparation is very important to find the lesion. Desirable bowel preparation drug must be clearly removed stool, effective on colonoscopic finding and pathologic finding, quickly administrated agent and eliminated stool, comfort for patient, and less side effects.

PEG is very safe osmotic laxative. New agent(coolprep) which add ascorbic acid is less salty and less volume. Picosulfate+magnesium citrate(picolyte) taste orange, can be easily prepared bowel for colonoscopy by good taste and small volume. Magnesium with citrate acts like osmotic agent, picosulfate acts irritant agent.

The investigators will compare with PEG+ascorbic acid and picosulfate+magnesium citrate about bowel preparation, patient's satisfaction, side effects to identify effectiveness of new bowel preparation drug.

ELIGIBILITY:
Inclusion Criteria:

* Age : over 19 years
* Who will be done colonoscopy
* Who accepted informed consent

Exclusion Criteria:

* Age : over 80 years
* Electrolyte imbalance
* Liver function test abnormality, ascites(over 2 times, >Child class B)
* ARF or CRF(GFS<30)
* Recent MI(< 6months) or Unstable angina pectoris
* Congestive heart failure(NYHA > 2)
* Inflammatory bowel disease
* Abdominal minor surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a total of 250 patients. All patient randomized PEG+ascorbica acid(coolprep) and picosulfate magnesium citrate(picolyte), each group will include 125 patients.
  The investigators decided sample size to 200 patients after comparing Ottawa scale. The investigators assumed there would be defference about 20 percent of bowel preparation between them. Recently, Ottawa scale of bowel preparation reported about 5 points. The investigators assumed that there could be differences between them about 1 point. The investigators decided each groups per 100 patients, if significance level was 0.05 and test power is 80 percent. The investigators start this study with a total of 220 patients because 10 percent of 200 patients could be drop out. The investigators readjust about 30 patients after interim analysis.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-06 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Ottawa scale | Ottawa scale will be checked at the end of the colonoscopy. Participants won't be followed up because of this study.
  * Ottawa scale
  Individual evaluation of right, mid, and left colon:
  No liquid - 0 Minimal liquid, no suctioning required - 1 Suction required to see mucosa - 2 Wash and suction - 3 Solid stool,not washable - 4
  Evaluation of the entire colon:
  Overall quantity of fluid 0-2 minimal -0 moderate - 1 Large - 2
  * Aronchick score scale Minimal liquid, visible more than 95% of colon mucosa - excellent Clear liquid covered 5~25% of mucosa, visible more than 90% of colon mucosa - good Solid stool, washable, visible more than 90% of colon mucosa - Fair Solid stool, not washable, visible less than 90% of colon mucosa not washable - Poor Bowel preparation is needed - Inadequate

SECONDARY OUTCOMES:
Patient satisfaction | Questionnaires related with satisfaction and side effects will be written just befor colonoscopy. Participants won't be followed up because of this study.
  Taste, Comfort
Symptoms related with bowel preparation | Questionnaires related with side effects will be written just befor colonoscopy. Participants won't be followed up because of this study.
  Nausea, Vomiting, Abdominal discomfort, Abdominal distension, Headache, Dizziness, Numbness

CONTACTS AND LOCATIONS:
Overall Officials: Jun Won Chung, Professor, Study Director — Gachon University Gil Medical School